CLINICAL TRIAL: NCT04201210
Title: A Phase II Stratified Trial to Assess Haploidentical T-depleted Stem Cell Transplantation in Patients With Sickle Cell Disease With no Available Sibling Donor
Brief Title: A Trial to Assess Haploidentical T-depleted Stem Cell Transplantation in Patients With SCD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Selim Corbacioglu, Head of the department, University of Regensburg
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-Haplo for SCD
Record Dates: First submitted 2019-12-02; First posted 2019-12-17 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: HbS Disease; Hemoglobin S Disease; Sickle Cell Anemia; Sickle Cell Disorders; Sickling Disorder Due to Hemoglobin S; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Patients who fulfill inclusion criteria will be stratified according to donor availability. Patients with a matched sibling donor (MSD; defined as 8/( or 10/10 allelic match) will be stratified into the control arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Patients with no matched sibling donor (MSD; defined as 8/( or 10/10 allelic match) will be stratified into the experimental arm
  Interventions: Other: TCRα/β+ and CD19+ depleted haploidentical stem cell transplantation
- Control Arm (Active Comparator): Patients with a matched sibling donor (MSD; defined as 8/( or 10/10 allelic match) will be stratified into the control arm
  Interventions: Other: Matched sibling donor transplantation

INTERVENTIONS:
Other: TCRα/β+ and CD19+ depleted haploidentical stem cell transplantation — Haploidentical 5+/10 HSCT from a relative, α/β T-depleted
  Arms: Experimental Arm
Other: Matched sibling donor transplantation — 10/10 HSCT - matched family donor
  Arms: Control Arm

SUMMARY:
HSCT is currently the only curative option for SCD but less than 20% of SCD patients have a MD donor available. So far, all curative approaches beyond a MSD HSCT at young age are non-satisfactory. With the lack of a suitable donor for the vast majority of patients, the major question of this trial is, if a haploidentical αß/CD19+ T-cell depleted HSCT can be a valid alternative to a MSD HSCT. The main challenge in non-malignant diseases is to offer a safe and GvHD-free HSCT without rejection.

DETAILED DESCRIPTION:
Can an α/ß depleted T-Haplo-HSCT with regard to disease free survival, adverse events and safety be considered equivalent to a matched sibling donor transplantation (MSD), in order to offer cure for the majority of patients with sickle cell disease.

The main questions of this trial are:

* Safety of a α/ß T-depleted haploidentical HSCT
* Incidence of acute and chronic GvHD
* Rate of rejection
* Immune reconstitution
* Fertility It is expected that the use of TCRαβ+ and CD19+ depleted haploidentical cell grafts in combination with the less aggressive and well tolerated conditioning regimen needed for patient preparation will be associated with a low risk of grade II-IV aGVHD and no extensive cGvHD, no graft failure and increase speed, spectrum and functionality of immune system reconstitution. This is supposed to reduce the incidence of severe infections leading to lower rates of transplantation related mortality (TRM).

ELIGIBILITY:
Inclusion Criteria:

* Age 2yrs to 35yrs
* Homozygous hemoglobin S disease or heterozygous hemoglobin SC or S 0/+
* Study specific consent given
* Preexisting severe or moderate SCD related complications:

  * Clinically significant neurological event (stroke) or deficit
  * Silent crisis, neurocognitive deficit
  * Pathological angio-MRI with TOF Sequence
  * TCD velocity >200 cm/s at 2 occasions >1 month apart
  * More than 5 vaso-occlusive crises (VOC) in the past 1 year or more than 20 VOC in a lifetime
  * Two or more episodes of acute chest syndrome (ACS) in a lifetime or one episode of ACS in the past 24 months
  * Chronic transfusion requirement or more than 8 transfusions or one exchange transfusion in a lifetime
  * Transfusion-refractory allo-immunization
  * More than five SCD-related hospitalizations in a lifetime
  * Beginning pulmonary hypertension
  * Osteonecrosis at more than 2 sites
  * Beginning SCD Nephropathy
  * Recurrent priapism (>2)

Exclusion Criteria:

* Karnofsky or Lansky Performance Score < 70%
* Patients with donor-specific antibodies (DSA) against the potential stem cell donor by either

  * Cell-based crossmatched assays (Complement-dependent cytotoxicity; CDC) or
  * Flow cytometry crossmatch test or
  * Solid-phase immunoassays (SPI) or
  * Modified SPI such as C4d and C1q assays Whichever method the participating center is experienced in.
* Patients with major AB0 incompatibility defined according to EBMT Handbook, Edition 2019 Tab 23.1.:

ABO incompatibility Recipient Donor Major O A O B O AB A AB B AB

* Cardiac function:

  * Ejection fraction at rest <45.0% on echocardiography or
  * Shortening fraction of <27.0% by echocardiogram or radionuclide scan (MUGA)
  * Patients with > grade II hypertension by Common Toxicity Criteria (CTC)
* Renal function:

  * Estimated creatinine clearance (for patients > 12 years) greater than 50.0 mL/minute
  * for pediatric patients (> 1 year to 12 years), GFR estimated by the updated Schwartz formula ≥ 90.0 mL/min/1.73 m2. If < 90 mL/min/1.73 m2, renal function must be measured by 24-hour creatinine clearance or nuclear GFR and must be > 70.0 mL/min/1.73 m2 or
  * Creatinine clearance below threshold defined for stem cell transplantation according to local clinical standard
* Pulmonary function:

  * DLCO >50% (adjusted for hemoglobin), and FVC and FEV1≥50%; children unable to perform for PFTs, O2 saturation <92% on room air.
* Liver function:

  * Total bilirubin > 2x the upper limit of normal (unless elevated bilirubin is attributed to Gilbert's Syndrome) and ALT/AST > 2.5x the upper limit of normal.
  * Chronic active viral hepatitis
* Women who are pregnant (positive serum or urine βHCG) or breastfeeding. Note: Women of childbearing potential must have a negative serum pregnancy test at study entry.
* Adults of reproductive potential not willing to use an effective method of birth control during study treatment and for at least 12 months thereafter,
* History of uncontrolled autoimmune disease or on active treatment
* Patient unable to comply with the treatment protocol
* Prior autologous or allogeneic hematopoietic stem cell transplant
* Vaccination with a live virus vaccine during the trial
* HIV infection
* Patients with a history of psychiatric illness or a condition which could interfere with their ability to understand the requirements of the study (this includes alcoholism/drug addiction)
* Patients unwilling or unable to comply with the protocol or unable to give informed consent.
* Concurrent severe or uncontrolled medical disease (e.g. uncontrolled diabetes, congestive heart failure, myocardial infarction within 6 months prior to the study, unstable and uncontrolled hypertension, chronic renal disease, or active uncontrolled infection) which by assessment of the treating physician could compromise participation in the study

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 212 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint: Composite Endpoint: Event free survival (EFS). | day 0 - day180
  Event is defined as incidence of acute GvHD (Grade III - IV), chronic GvHD (moderate/severe), graft failure (GF), or death (from any reason).

SECONDARY OUTCOMES:
Overall survival | up to 2 years after transplantation
  Overall survival rate (OS) is defined as time from transplantation to death or last follow-up and will be assessed at Day 100 and after 1 year and 2 years.
Disease free survival | up to 2 years after transplantation
  • Disease-free survival (DFS) is defined as the minimum time to recurrence, to death or to the last follow-up, from the time of transplantation and will be assessed at Day 100 and after 1 year and 2 years.
Graft failure | up to 2 years after transplantation
  defined as initial neutrophil engraftment followed by a decline in ANC <500/µl that is unresponsive to growth factor therapy and/or other intervention
Quality of life: EQ-5D | up to 2 years after transplantation
  Adult patients ≥18 years. The European Quality of Life 5 Dimension (EQ-5D) questionnaire has two components: health state description and evaluation.
  In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are.
Quality of life: PedsQL | up to 2 years after transplantation
  The Pediatric Quality of Life Inventory (PedsQL) is a 23-item generic health status instrument with parent and child forms that assesses five domains of health (physical functioning, emotional functioning, psychosocial functioning, social functioning, and school functioning) in children and adolescents ages 2 to 18.
Quality of life: FACT-BMT | up to 2 years after transplantation
  Functional Assessment of Cancer Therapy-Bone Marrow Transplant (adult patients ≥18 years). FACT-BMT form was designed to measure the QoL in patients undergoing bone marrow transplantation. It combines the FACT-G, an assessment of physical well-being, social/family well-being, emotional well-being and functional well-being, with Bone Marrow Transplantation Sub-scale(BMTS) to measure the QOL of BMT patients.

CONTACTS AND LOCATIONS:
Overall Officials: Selim Corbacioglu, MD, Principal Investigator — University Hospital of Regensburg
Locations (9):
- St. Anna Kinderspital, Vienna, Austria
- Germany (8):
  - University Hospital Aachen, Children's Hospital, Aachen
  - Charité University medicine, Clinic for Hematology, Oncology, Berlin
  - University Hospital Duesseldorf, Clinic for Pediatric Oncology, - Hemtaology and Clinical Immunology, Düsseldorf
  - University Hospital of Frankfurt, Clinic for Paediatrics and Adolescent Medicine, Frankfurt
  - University Hospital Heidelberg, Department of Pediatric Hematology, Oncology and Immunology, Heidelberg
  - University Hospital Regensburg, Dept. of Ped. Hematology, Oncology and Stem Cell Transplantation, Regensburg
  - University Children's Hospital Tübingen, Tübingen
  - University Children's Hospital Würzburg, Würzburg